CLINICAL TRIAL: NCT06832540
Title: Mass Balance Study of [14C] TJ0113 in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou PhecdaMed Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJJS01-002
Record Dates: First submitted 2025-02-06; First posted 2025-02-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy Chinese Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]TJ0113 (Experimental): A single oral dose of approximately 200 mg/100 μCi of the oral formulation of [14C] TJ0113
  Interventions: Drug: [14C]TJ0113

INTERVENTIONS:
Drug: [14C]TJ0113 — Subjects will receive a single oral dose of approximately 200 mg/100 μCi of the oral formulation of [14C] TJ0113 under fasted conditions.

SUMMARY:
Mass Balance Study of [14C] TJ0113 in Healthy Chinese Subjects

DETAILED DESCRIPTION:
This is a single-center, single-dose and open-label trial designed to enroll 6-8 healthy adult male subjects to evaluate the mass balance of [14C]TJ0113 in these subjects. Each subject will receive a single oral dose of approximately 200 mg /100 μCi [14C]TJ0113 oral formulation; after administration, blood, urine, and stool samples will be collected at specified time points/intervals during the study. The total radioactivity in whole blood and plasma, as well as the plasma concentrations of TJ0113 and its metabolites will be determined to calculate the pharmacokinetic (PK) parameters of [14C]TJ0113 and its metabolites in plasma and whole blood as well as the PK parameters of TJ0113 and its metabolites in plasma, and to understand the distribution of total radioactivity in whole blood and plasma; the radioactivity in urine and feces will be determined to obtain the data on total recovery, excretion and main routes of excretion; the metabolic pathways of TJ0113 in humans will be determined through radiolabeled metabolite profiling and structural identification of major metabolites in plasma, urine, and feces.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese males;
2. Age at informed consent: 18-45 years (inclusive);
3. Body mass index (BMI) ranging from 19 to 26 kg/m2 (inclusive) and body weight ≥ 50 kg;
4. Fully understand the objectives and requirements of this study, and voluntarily sign the informed consent form;
5. Able to communicate well with study personnel and complete the study according to the protocol.

Exclusion Criteria:

Auxiliary examination:

1. Subjects who have abnormal and clinically significant results of comprehensive physical examination, digital anal examination, laboratory tests (hematology, blood chemistry, coagulation function, urinalysis, stool routine + occult blood, thyroid function), 12-lead ECG, ophthalmic examination (slit-lamp, intraocular pressure and fundus radiography), chest X-ray (anteroposterior) and abdominal B ultrasound (liver, gallbladder, pancreas, spleen and kidney);
2. Subjects with unqualified vital signs that remain unqualified upon retesting;
3. Subjects who have a resting corrected QT interval (QTcF) > 450 ms (corrected according to Fridericia's formula) or QRS > 120 ms as determined by 12-lead electrocardiogram (ECG), or a previous history of long QT syndrome;
4. Subjects who have any clinically significant abnormality in hepatitis B surface antigen, hepatitis B E antigen, hepatitis C virus antibody (anti-HCV), treponema pallidum antibody test, and human immunodeficiency virus antibody (anti-HIV) as judged by the investigator;

   Medication History:
5. Subjects who use any drug inhibiting or inducing hepatic drug-metabolizing enzyme activity (see Appendix 1 for details) within 30 days before screening;
6. Subjects who use any prescription drugs, over-the-counter drugs, Chinese herbal medicines and food supplements (such as vitamins and calcium supplements) from 14 days before screening to predose;

   Disease and Surgical History:
7. Subjects who have febrile illness or active infection within 14 days before screening;
8. Subjects who have gastrointestinal diseases causing clinically significant symptoms such as nausea, vomiting, diarrhea or malabsorption syndrome, or a history of severe vomiting or diarrhea within one week before screening;
9. Subjects who have a history of any clinically significant disease or any disease or condition that may affect the study results in the opinion of the investigator, including but not limited to cardiovascular system, respiratory system, endocrine system, nervous system, digestive system, urinary system or blood, immune, mental and metabolic diseases;
10. Subjects who have dysphagia or any condition that may affect oral administration and drug absorption (e.g., cholecystectomy, gastric bypass, duodenotomy, colectomy, post-gastrointestinal resection, ulcerative colitis, symptomatic/inflammatory bowel disease, intestinal obstruction, etc.);
11. Subjects who have undergone major surgery within 6 months before screening or have incomplete healing of surgical incision, including but not limited to any surgery with significant bleeding risk, prolonged general anesthesia, or incisional biopsy or significant traumatic injury; or who have undergone surgery affecting drug absorption, distribution, metabolism, excretion, or plan to undergo surgery during the study period;
12. Subjects who have drug, environmental, food allergy or allergic constitution, or may be allergic to the investigational product judged by the investigator;
13. Subjects who have hemorrhoids or perianal diseases accompanied by regular/ongoing hematochezia, irritable bowel syndrome, inflammatory bowel disease;

    Life Style:
14. Habitual constipation or diarrhea;
15. Subjects who have alcoholism or regular drink within 6 months before screening, defined as drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits 40% or 150 mL of wine), or have a breathalyzer test result > 0 mg/100 ml at screening, or unable to abstain from alcohol during the study;
16. Subjects who smoke more than 5 cigarettes per day or habitually use nicotine-containing products within 3 months before screening, or inability to abstain during the study;
17. Subjects who abuse drugs or use soft drugs (such as marijuana) 3 months before screening or take hard drugs (such as amphetamines, phencyclidine, etc.) 1 year before screening; or have positive urine drug test during screening;
18. Subjects who have special requirements for diet or fail to follow the standard diet (such as intolerant of standard meals); habitually drink grapefruit juice or excessive tea, coffee and/or caffeine beverages, or unable to abstain during the study; refuse to discontinue any beverages containing xanthine derivatives, such as caffeine (coffee, tea, cola, chocolate, etc.) from 48 hours pre-dose until the end of the study; refuse to discontinue animals' viscera, seafood, soy products and other foods containing high purine;
19. Subjects who have strenuous exercise or other factors affecting drug absorption, distribution, metabolism and excretion;
20. Lactose intolerance (subjects who have had diarrhea from drinking milk);

    Others:
21. Subjects who are exposed to radioactivity for a prolonged period, or have significant radiation exposure (≥ 2 chest/abdominal CT scans, or ≥ 3 other X-ray examinations) within one year before screening, or have participated in radiopharmaceutical labeling trials within one year before screening;
22. Subjects who have a history of syncope due to the needles or blood, or difficult blood collection or cannot tolerate venipuncture for blood collection;
23. Subjects who have participated in any clinical trial within 3 months before screening and have received an investigational product or used an investigational device; or those who plan to participate in other clinical trials during this study, or subjects who do not participate in the clinical trial in person;
24. Subjects who have been vaccinated within 1 month before screening or planned to receive vaccination during the study;
25. Subjects who plan to father a child or donate sperm from the time of signing the informed consent form to 1 year after completing the study, or do not agree to take strict contraceptive measures (see Appendix 3 for details) for themselves and their spouses from the time of signing the informed consent form to 1 year after completing the study;
26. Subjects who have blood loss or blood donation ≥ 400 mL within 3 months before screening, or blood transfusion or blood component within 1 month before screening, or blood donor during planned medication and within 3 months after discontinuation;
27. Subjects who have any other factor that the investigator considers inappropriate for participation in this study or the subject withdraws from the study for his/her own reasons.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
The excretion ratio of total radioactivity at each time interval and the cumulative recovery of total radioactivity in urine and feces | Predose up to 240 hours after administration of [14C]TJ0113
  The excretion ratio of total radioactivity at each time interval and the cumulative recovery of total radioactivity in urine and feces
Pharmacokinetic parameters of total radioactivity in plasma: Cmax | Predose up to 168 hours after administration of [14C]TJ0113
  Maximum concentration
Pharmacokinetic parameters of total radioactivity in plasma: Tmax | Predose up to 168 hours after administration of [14C]TJ0113
  Time to Maximum Concentration
Pharmacokinetic parameters of total radioactivity in plasma: t1/2 | Predose up to 168 hours after administration of [14C]TJ0113
  Half Life
Pharmacokinetic parameters of total radioactivity in plasma: MRT | Predose up to 168 hours after administration of [14C]TJ0113
  Mean Residence Time
Pharmacokinetic parameters of total radioactivity in plasma: AUC | Predose up to 168 hours after administration of [14C]TJ0113
  Area Under the Plasma Concentration-time Curve

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No